CLINICAL TRIAL: NCT00159718
Title: Double Blind Atorvastatin Amlodipine Study (DUAAL) Effect Of Amlodipine, Atorvastatin And The Combination On Transient Myocardia Ischemia In Coronary Artery Disease.
Brief Title: Double Blind Atorvastatin Amlodipine Study
Acronym: DUAAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0531031
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Angina
MeSH Terms: conditions — Angina Pectoris | interventions — Amlodipine; Atorvastatin

INTERVENTIONS:
Drug: amlodipine
Drug: atorvastatin

SUMMARY:
To evaluate and compare the safety and efficacy of amlodipine, atorvastatin and the combination in patients with symptomatic myocardial ischemia.

Amlodipine's use in angina has been well documented in clinical trials such as the Circadian Anti-Ischemia Program in Europe (CAPE), but the impact on vascular inflammation in clinical practice has not been tested. Furthermore, the potentially synergistic benefit of atorvastatin and amlodipine on inflammation ischemic activity has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Holter monitoring at baseline which demonstrates a total of 15 minutes of ischemia and/or 3 ischemic events per 48 hours.
* Total cholesterol > 5.2 mmol/L (200 mg/dL) on diet alone.

Exclusion Criteria:

* Myocardial infarction within 2 months prior to the study.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2001-07; Study Completion 2007-01

PRIMARY OUTCOMES:
From the 48 hour holter monitoring the number of ischemic episodes will be assessed at baseline (week 1), week 18 and at the final visit (week 26).

SECONDARY OUTCOMES:
Inflammatory markers will be assessed at baseline (week 2), week 6, week 18 and
week 26. Inflammatory markers to be analyzed are the following: C-reactive
protein, amyloid A and interleukin 6.
From the exercise tolerance tests the time to onset of 1 mm ST depression, time to
onset of angina and total exercise time will be assessed at baseline (week 2),
week 18 and week 26.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Croatia (2):
  - Pfizer Investigational Site, Rijeka
  - Pfizer Investigational Site, Zagreb
- Czechia (5):
  - Pfizer Investigational Site, Ostrava-Kunčice
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Příbram
  - Pfizer Investigational Site, Rokycany
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Hungary (5):
  - Pfizer Investigational Site, Debrecen, Budapest
  - Pfizer Investigational Site, Balatonfüred
  - Pfizer Investigational Site, Berettyóújfalu
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Zalaegerszeg
- Latvia (3):
  - Pfizer Investigational Site, Daugavpils
  - Pfizer Investigational Site, Riga
  - Pfizer Investigational Site, Valmiera
- Norway (2):
  - Pfizer Investigational Site, Baerum Postterminal
  - Pfizer Investigational Site, Oslo
- Poland (4):
  - Pfizer Investigational Site, Bytom
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Warsaw
- Romania (3):
  - Pfizer Investigational Site, Brasov, Jud. Brasov
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Craiova
- Pfizer Investigational Site, Bratislava, Slovakia
- South Africa (2):
  - Pfizer Investigational Site, Observatory, CAPE
  - Pfizer Investigational Site, Parow, CAPE
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Çapa, Istanbul
  - Pfizer Investigational Site, Bornova/izmir
  - Pfizer Investigational Site, Samsun
- Pfizer Investigational Site

REFERENCES:
- [Derived] Deanfield JE, Sellier P, Thaulow E, Bultas J, Yunis C, Shi H, Buch J, Beckerman B. Potent anti-ischaemic effects of statins in chronic stable angina: incremental benefit beyond lipid lowering? Eur Heart J. 2010 Nov;31(21):2650-9. doi: 10.1093/eurheartj/ehq133. Epub 2010 May 21. PMID 20494902
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531031&StudyName=Double+Blind+Atorvastatin+Amlodipine+Study+%28DUAAL+Study%29+